CLINICAL TRIAL: NCT00304304
Title: Community - Based Asthma Intervention in Subsidized Preschools
Brief Title: HealthSpark 2: Improving Asthma Care for Preschool Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: Health Foundation of South Florida (Other); Ounce of Prevention Fund (Other); The Early Childhood Initiative Foundation (Other)
Responsible Party: Principal Investigator, Jeffrey P. Brosco, Professor, Clinical Pediatrics, University of Miami
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: 20057395
Record Dates: First submitted 2006-03-16; First posted 2006-03-17 (Estimated); Last update posted 2016-02-17 (Estimated); Status verified 2016-02

CONDITIONS: Asthma
Keywords: child care centers; asthma triggers; community-based research
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention - asthma education (Active Comparator): CCC received asthma education in the first 6 months of the study
  Interventions: Behavioral: Asthma education
- Wait-list control (Placebo Comparator): CCC received asthma education in second 6 months of study
  Interventions: Behavioral: Asthma education

INTERVENTIONS:
Behavioral: Asthma education — Research assistant worked with CCC staff on asthma prevention

SUMMARY:
From a previous community needs survey, we determined that asthma was a particular problem in our community-based research network of child care centers. This study will examine whether a moderate intervention can help these centers improve their "asthma-friendly" rating as per NHLBI guidelines. We will both center directors and parents to establish baseline data on child health and the "asthma-friendliness" of each center. We will use a wait-list control, with all centers eventually receiving the intervention.

DETAILED DESCRIPTION:
Asthma is the most common chronic health problem affecting children in the U.S., and it is getting worse. Children under the age of 18 years account for one third of the nation's asthma sufferers. The percent of children with asthma has increased from 3% in 1981 to 6% in 2003. Asthma is a leading reason for hospitalizations of children under the age of 15 years and causes 14 million days of missed school each year. Previous studies suggest particularly high asthma rates among Hispanic and African-American populations. Poverty, increased exposure to indoor allergens, low education level, poor access to healthcare, and failure to take prescribed medicines increase the likelihood of having a severe asthma attack, or dying of asthma.

According to the results of HealthSpark I, children in the target communities have rates of asthma that are more than three times the national average. 29.3% of HealthSpark families with children ages 3 to 5 years responded "yes" to the question, "Did a doctor ever tell you that your child has asthma?" In a national survey in 2002, only 7.3% of parents with children ages 0 to 4 years responded "yes" to the same question. The high rate of asthma among HealthSpark families is similar to recent reports of high prevalence in Harlem, NY, and other underserved, minority communities.

Of HealthSpark parents reporting that their child has asthma, 38.7% also reported that their child was taking a medication regularly for more than a year. It is reasonable to assume that most of these were asthma medications, which suggests that approximately 11.3% of the total HealthSpark population has moderate to severe asthma. These children also had high rates of comorbidity. HealthSpark children with asthma were twice as likely as children without asthma to be limited in their daily activities, and three times as likely to require increased medical, educational, and mental health services. HealthSpark children with asthma were also two to three times as likely than children without asthma to have early signs of attention deficit hyperactivity disorder (ADHD).

Our analysis also revealed ethnic differences in asthma prevalence consistent with national patterns. African American children were nearly twice as likely to have a diagnosis of asthma when compared with Hispanic children (40.6% vs. 23%). None of these findings were related to access to child health care. Children with asthma, in fact, had better access to care than children without asthma, as demonstrated by the following measures: having a regular source of care (99.4% vs 91%), having health insurance (92.5% vs. 88.6%), and having a regular doctor that their parents could name (94.0% vs. 86.5%). Children with moderate/severe asthma had even better access to care: 98.4% of parents could name their physician and 97% had health insurance for their child.

In 1989, the National Asthma Education and Prevention Program (NAEPP) was initiated by the National Heart, Lung, and Blood Institute (part of the NIH) to address the growing problem of asthma in the United States. To accomplish these broad program goals, the NAEPP works with intermediaries including major medical associations, voluntary health organizations, and community programs to educate patients, health professionals, and the public. The ultimate goal of the NAEPP is to enhance the quality of life for patients with asthma and decrease asthma-related morbidity and mortality. As part of this broad program, the NHLBI released guidelines for CCCs to provide optimal care for children with asthma. These "asthma-friendly" guidelines are at the core of this proposal.

This project is a community-based intervention to begin to improve asthma care among these preschool children. The target population is 2000 children aged 1-5 years who attend the 51 child care centers that remain as part of the SPARK network.

The long-term goals of this project are to (a) improve the health of children by improving asthma care in the targeted, underserved areas of Miami-Dade County and (b) to enhance readiness for school by reducing the burden of asthma and related conditions.

The specific objectives for this project are:

1. Document the prevalence, severity, and impact of asthma among preschool children attending the 51 SPARK child care centers (CCCs) in Allapatah/Model City and Homestead/Florida City.
2. Identify barriers to optimal asthma care in these children.
3. Determine how "asthma-friendly" each child care center is according to guidelines of the National Heart, Lung, and Blood Institute (part of the NIH) (see Appendix I).
4. Work with CCCs and community health clinics to improve clinical outcomes for children with asthma.

Outcomes

1. We will better understand the prevalence, severity, and impact of asthma among preschool children in underserved communities (parent surveys).
2. We will identify barriers to optimal, community-based asthma care projects (parent surveys and CCC survey).
3. We will increase the number of CCCs that are "asthma-friendly" (CCC surveys, site visit).
4. We will improve clinical outcomes for children with asthma (parent survey).
5. We will increase the number of children with written asthma plans from an estimated 10% to greater than 50%.

Other outcomes:

Baseline correlations to identify significant relationships among individual characteristics including asthma severity, healthcare utilization, healthcare access, comorbidity, quality of life, environmental exposures, maternal health literacy, and maternal education

ELIGIBILITY:
Inclusion Criteria:

* Children ages 1 - 5 years, enrolled in one of the designated SPARK child care centers

Exclusion Criteria:

* Children under the age of 1 year
* Children whose parents do not want to participate
* Children whose child care centers do not want to participate

Ages: 1 Year to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 2000 (Actual)
Dates: Start 2006-02; Primary Completion 2006-12 (Actual); Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
6 month post-intervention: quality of CCC asthma policy | 6 months
  Did CCC have appropriate policy

SECONDARY OUTCOMES:
6 month post-intervention changes in asthma outcomes | 6 months
  Parent-report of fewer asthma symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey P Brosco, MD PhD, Principal Investigator — University of Miami
Locations (1):
- University of Miami Mailman Center for Child Development, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No